CLINICAL TRIAL: NCT04517071
Title: Predictors of Success Following Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Other Study IDs: 9700778J
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2018-10

CONDITIONS: Focus of Study is Patient Responses to an Obesity Management Questionnaire Administered by SGH Life Centre

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to consolidate the contributions of various medical, social and psychological predictors of success following bariatric surgery amongst Singaporeans.

ELIGIBILITY:
Inclusion Criteria:

* Undergone bariatric surgery within SGH lIfe centre and must have completed the intake questionnaire.

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Singaporeans who have undergone bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Weight Loss | Immediately post-surgery within first year
  Weight Loss in Kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No